CLINICAL TRIAL: NCT00082251
Title: Safety & Efficacy of a Combination Niacin ER/Simvastatin in Patients With Dyslipidemia: A Dose-Ranging Study - SEACOAST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kos Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 019-01-03-CR; SEACOAST
Record Dates: First submitted 2004-05-03; First posted 2004-05-05 (Estimated); Last update posted 2006-11-01 (Estimated); Status verified 2006-10

CONDITIONS: Hypercholesterolemia
Keywords: Dyslipidemia; High Blood Cholesterol; Coronary Heart Disease; Hypertension; National Cholesterol Education Program; Adult Treatment Panel III; Niacin; Simvastatin; Diabetes; Peripheral Vascular Disease; Cerebrovascular disease; Stroke; High-Density Lipoprotein Cholesterol; Hydroxymethyl Glutaryl Coenzyme A; High-Sensitivity C-Reactive Protein; Low-Density Lipoprotein Cholesterol; Lipoprotein (a); Lipoprotein A-I; Total Cholesterol; Triglycerides
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias; Coronary Disease; Hypertension; Diabetes Mellitus; Peripheral Vascular Diseases; Cerebrovascular Disorders; Stroke | interventions — Simvastatin

INTERVENTIONS:
Drug: Niacin extended release and simvastatin tablets

SUMMARY:
The purpose of this study is to compare the effectiveness and safety of different doses of Niacin ER/Simvastatin (NS), in subjects with elevated fat levels in their blood (dyslipidemia).

DETAILED DESCRIPTION:
The purpose of this study is to compare the efficacy and safety of different doses of Niacin ER/Simvastatin (NS), in subjects with elevated fat levels in their blood (dyslipidemia).

ELIGIBILITY:
Inclusion Criteria:

* Patient has primary Type II hyperlipidemia or mixed dyslipidemia
* If the patient is currently taking anti-dyslipidemic medications other than Zocor, he/she is willing to withdraw from these medications
* Reasonable compliance with a standard cholesterol-lowering diet for a minimum of 4 weeks prior to screening and for the duration of the study.
* LDL-C levels and/or Non HDL-C levels above normal for patients

This study will be conducted both in the USA and internationally.

Exclusion Criteria:

* Patient has an allergy, hypersensitivity, or intolerance to niacin, statins, or their derivatives
* HbA1c ≥ 9% in diabetic patients

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

REFERENCES:
- [Background] National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). Third Report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III) final report. Circulation. 2002 Dec 17;106(25):3143-421. No abstract available. PMID 12485966
- [Background] Grundy SM, Cleeman JI, Merz CN, Brewer HB Jr, Clark LT, Hunninghake DB, Pasternak RC, Smith SC Jr, Stone NJ; National Heart, Lung, and Blood Institute; American College of Cardiology Foundation; American Heart Association. Implications of recent clinical trials for the National Cholesterol Education Program Adult Treatment Panel III guidelines. Circulation. 2004 Jul 13;110(2):227-39. doi: 10.1161/01.CIR.0000133317.49796.0E. PMID 15249516
- [Background] Cui Y, Blumenthal RS, Flaws JA, Whiteman MK, Langenberg P, Bachorik PS, Bush TL. Non-high-density lipoprotein cholesterol level as a predictor of cardiovascular disease mortality. Arch Intern Med. 2001 Jun 11;161(11):1413-9. doi: 10.1001/archinte.161.11.1413. PMID 11386890
- [Background] Bittner V, Hardison R, Kelsey SF, Weiner BH, Jacobs AK, Sopko G; Bypass Angioplasty Revascularization Investigation. Non-high-density lipoprotein cholesterol levels predict five-year outcome in the Bypass Angioplasty Revascularization Investigation (BARI). Circulation. 2002 Nov 12;106(20):2537-42. doi: 10.1161/01.cir.0000038496.57570.06. PMID 12427648
- [Background] Marcelino JJ, Feingold KR. Inadequate treatment with HMG-CoA reductase inhibitors by health care providers. Am J Med. 1996 Jun;100(6):605-10. doi: 10.1016/s0002-9343(96)00011-3. PMID 8678079
- [Background] Pearson TA, Laurora I, Chu H, Kafonek S. The lipid treatment assessment project (L-TAP): a multicenter survey to evaluate the percentages of dyslipidemic patients receiving lipid-lowering therapy and achieving low-density lipoprotein cholesterol goals. Arch Intern Med. 2000 Feb 28;160(4):459-67. doi: 10.1001/archinte.160.4.459. PMID 10695686
- [Background] Mosca L, Grundy SM, Judelson D, King K, Limacher M, Oparil S, Pasternak R, Pearson TA, Redberg RF, Smith SC Jr, Winston M, Zinberg S. AHA/ACC scientific statement: consensus panel statement. Guide to preventive cardiology for women. American Heart Association/American College of Cardiology. J Am Coll Cardiol. 1999 May;33(6):1751-5. doi: 10.1016/s0735-1097(99)00190-4. No abstract available. PMID 10334455
- [Background] Guyton JR, Goldberg AC, Kreisberg RA, Sprecher DL, Superko HR, O'Connor CM. Effectiveness of once-nightly dosing of extended-release niacin alone and in combination for hypercholesterolemia. Am J Cardiol. 1998 Sep 15;82(6):737-43. doi: 10.1016/s0002-9149(98)00448-2. PMID 9761083
- [Background] Reaven P, Witztum JL. Lovastatin, nicotinic acid, and rhabdomyolysis. Ann Intern Med. 1988 Oct 1;109(7):597-8. doi: 10.7326/0003-4819-109-7-597_2. No abstract available. PMID 3421570
- [Background] Norman DJ, Illingworth DR, Munson J, Hosenpud J. Myolysis and acute renal failure in a heart-transplant recipient receiving lovastatin. N Engl J Med. 1988 Jan 7;318(1):46-7. doi: 10.1056/NEJM198801073180110. No abstract available. PMID 3275891